CLINICAL TRIAL: NCT07293364
Title: A Prospective, Open- Label, Single-country (Algeria), Interventional Study to Assess Measurements of Functional C1-inhibitor Alone for Hereditary Angioedema Diagnosis: The AHAE Study
Brief Title: A Study to Learn About the C1-Inhibitor Function as Diagnosis for Hereditary Angioedema
Acronym: AHAE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: CRO Axelys Santé DZ (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TAK-743-4028
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspected HAE Participants (Experimental): Participants with suspected HAE having a high suspicion of bradykinin-mediated HAE (no urticaria or itching, lasting between 1 and 5 days, non-responsive to antihistamine and corticosteroid treatments) and/or family members of known HAE participants will be enrolled in the study.
  Interventions: Diagnostic Test: Technochrom C1-INH Kit

INTERVENTIONS:
Diagnostic Test: Technochrom C1-INH Kit — HAE biological diagnostic test that uses functional C1-INH technique by colorimetric method versus the reference test defined as the SoC (C4 and C1-INH antigenic level measurement and functional C1-INH assay).

SUMMARY:
Hereditary angioedema (HAE) is a rare condition. It causes sudden swelling under the skin and inside the body, like in the belly, throat, or genitals. This swelling happens because of a temporary leak in blood vessels but does not cause itching or hives. HAE is classified based on the amount of a protein in the blood called C1-inhibitor (C1INH): HAE with normal C1INH levels and function (HAE-nC1INH) and HAE with deficiency in C1INH levels (HAE-C1INH-Type1) or dysfunction (HAE-C1INH-Type2). This study will focus on the practical use and accuracy of measuring the C1INH function alone to diagnose HAE-C1INH-Type1 and HAE-C1INH-Type2 compared to the tests used in normal clinical practice in Algeria.

The main goal of the study is to see how well a test focusing on the C1INH function alone works to diagnose HAE-C1INH as compared to the tests used in normal clinical practice (standard of care or SoC) in Algeria. Another aim is to determine a reference value (helps in determining the accuracy) of the C1INH function test. This study will also help to find out how many people who are thought to have HAE or who have family members with HAE actually get diagnosed and to gather participants' health background information, such as their age when they were diagnosed, what signs and symptoms they had, how long it took to get diagnosed, and how they were sent to the doctors or specialists who treated them.

During the study all participants will undergo two different methods of HAE testing: the test focusing on the C1INH function alone and the SoC tests. Test results will be confirmed via a second test run for newly index cases or for discordant results, but participants with a test result of "no HAE" and positive cases recruited through family screening will not undergo a second confirmatory test. In case of discordant test results in the second round, participants will undergo a third confirmatory test round. Participants can visit the clinic up to three times during the study. No further follow up is planned for participants, even for those who are diagnosed with HAE.

ELIGIBILITY:
Inclusion Criteria

1. Adult and pediatric participants of both sexes (children over the age of 12 years).
2. Participants providing a signed informed consent form (ICF), or parental consent for minors.
3. Participants should also meet one of the 2 inclusion criteria below:

   1. Participants with a high suspicion of bradykinin-mediated HAE, referred to the center. This includes recurrent episodes of nonpitting angioedema without urticaria or itching, lasting between 1 and 5 days, and non-responsive to antihistamine and corticosteroid treatments.
   2. Family members (from 1st to 4th degree relatives) of known HAE participants.

Exclusion Criteria

1. Confirmed diagnosis of HAE-C1INH-Type1 or HAE-C1INH-Type2.
2. Angioedema with urticaria or itching (suggesting histaminergic etiology).
3. Angioedema episodes lasting less than (<)1 day or greater than (>)5 days (not consistent with bradykinin-mediated HAE).
4. Any condition deemed unsuitable by the investigator that may interfere with study procedures or data integrity.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-01-07 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Technochrom Compared to Standard of Care (SoC) for HAE Diagnosis | Up to 12 months
  The diagnostic accuracy of isolated functional C1-inhibitor (C1-INH) measurement using Technochrom C1-INH kits, compared to the SoC (McNemar's test) as confirmatory testing for HAE diagnosis will be reported.

SECONDARY OUTCOMES:
Laboratory-specific Cut-off Values for Functional C1-INH Measurement Using Technochrom | Up to 12 months
  Laboratory-specific cut-off values for functional C1-INH measurement in the Algerian population using the Technochrom C1-INH kit and assess their impact on diagnostic accuracy will be reported.
Sensitivity and Specificity of Technochrom Compared to Isolated Complement Component Test (C4 assay) for HAE Detection | Up to 12 months
  Sensitivity and specificity of Technochrom compared to isolated C4 assay will be evaluated.
Likelihood Ratios of Technochrom Compared to Isolated C4 Assay for HAE Detection | Up to 12 months
  Positive and negative likelihood ratios of the Technochrom compared to isolated measurement of antigenic C4 assay will be evaluated.
Sensitivity and Specificity of Technochrom Compared to C4 Assay and C1-INH Antigenic Testing | Up to 12 months
  Sensitivity and specificity of Technochrom compared to C4 assay and C1-INH antigenic testing will be evaluated.
Likelihood Ratios of Technochrom Compared to C4 Assay and C1-INH Antigenic Testing | Up to 12 months
  Positive and negative likelihood ratios of the Technochrom compared to C4 and C1-INH antigenic testing will be evaluated.
Diagnostic Performance of Technochrom in Detecting Functional C1-INH Deficiency and its Impact on Accuracy and Reliability in Clinical Practice | Up to 12 months
  Diagnostic performance assessment of Technochrom in detecting functional C1-INH deficiency, including its potential to enhance accuracy and reliability in clinical practice will be reported.
Number of Participants Categorized by Their Epidemiological, Clinical and Biological Characteristics | Up to 12 months
  Epidemiological, clinical, and biological characteristics of participants, including age at diagnosis, clinical presentation, diagnostic delay, and referral pathways will be reported.
Diagnostic Rate of Functional C1-INH Deficiency Using Technochrom in Highly Suspected Participants and Family Screening | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- EPH de Rouiba (Etablissement Public Hospitalier), Algiers, Algeria

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/e5ca430010de408c??page=1&idFilter=TAK-743-4028